CLINICAL TRIAL: NCT04337411
Title: Do Time-related Trajectories of Muscle Alterations Predict Gait Recovery in Acute Stroke Patients? A Study Protocol for Two Cohort Studies
Brief Title: Muscle Trajectories in Acute Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Lotte Cuypers, Doctoral Researcher, Vrije Universiteit Brussel
Other Study IDs: Muscle trajectories
Record Dates: First submitted 2020-03-20; First posted 2020-04-07 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Stroke
Keywords: Stroke; Acute; Subacute; Muscle; Inflammation; Gait; Sarcopenia
MeSH Terms: conditions — Stroke; Inflammation; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Non-ambulatory acute stroke survivors at admission (Functional Ambulation Categories (FAC) ≤ 2)
  Interventions: Other: Follow-up assessments
- Cohort 2: Ambulatory acute stroke survivors at admission (Functional Ambulation Categories (FAC) ≥ 3)
  Interventions: Other: Follow-up assessments

INTERVENTIONS:
Other: Follow-up assessments — Longitudinal evaluation of recovery

SUMMARY:
The aim of this study is to explore time-related trajectories of muscle alterations and inflammation in acute hospitalized stroke patients. Furthermore, the researchers want to gain insight in the predictive values of these time-related trajectories towards gait recovery in the acute stroke population.

DETAILED DESCRIPTION:
STUDY DESIGN:

Two longitudinal prospective cohort studies will be conducted in which non-ambulatory (cohort 1) and ambulatory (cohort 2) acute stroke patients will participate.

PATIENT RECRUITMENT:

The investigators aim to recruit 200 subjects (100/cohort). Patients will be recruited at the Neurology ward of the UZ Brussel.

PROCEDURE:

All stroke survivors admitted to the Neurology ward of UZ Brussel will be screened for eligibility. Afterwards, an informed consent will be conducted for all subjects who met the inclusion criteria.

Baseline assessments (T0) of gait recovery outcomes on the one hand and predictors for gait recovery on the other hand will be measured. To predict gait recovery, researchers will observe two novel biomarkers: stroke-induced muscle wasting and inflammation. Furthermore, the investigators will also assess relevant known predictors for gait recovery to compare the relevance of the novel markers. T0 assessments will start preferably within 3 days post-stroke.

To assess time-related trajectories of muscle alterations and inflammation, follow-up assessments of these predictors will be performed 3 days after baseline assessments (T1), at discharge (T2) and 3 months follow-up (T3). T1 follow-up measurements will only be possible for patients with motor impairments post-stroke since they have a longer stay at the hospital compared to patients without motor impairments after stroke (mean hospital stay of 5 to 8 days for patients without or with motor impairments post-stroke respectively).

The assessments of the gait recovery outcome measures will be repeated at discharge (T2) and 3 months follow-up (T3).

MATERIALS:

To measure gait recovery in acute stroke survivors, the researchers will make use of wearable gait sensors (Physiolog®, Gait Up SA, Switzerland) to register gait speed and a lightweight chest carrying gas analysis system (Metamax 3B, Cortex, Germany) to measure cardiorespiratory parameters.

For the predictors, investigators will use handheld dynamometers (MicroFET2 and Martin Vigorimeter) to assess muscle strength, grip strength and muscle fatigue. Furthermore, researchers need a Bioelectrical Impedance analysis (BIA) device (Bodystat® QuadScan 4000, UK) to assess the muscle mass of our subjects and a portable ultrasound system (Viamo SV 7 with linear-array transducer, Canon Medical Systems, Netherlands) to assess muscle architecture.

STATISTICAL ANALYSIS:

Various biomarkers will be observed at each of the planned time points. Because the aim is to make correct predictions based on any information that is available at the early stages, the observations will not only be considered as such, but also summarized in terms of their time- related characteristics, such as steepest drop, frequency of improvement, or any other characteristic that may reveal itself as distinguishing. These predictors will be combined into predictive models such as random forests and boosting to establish the best combinations for making good predictions while accommodating inter-predictor correlations. The quality of the models will be established with cross-validation. The large set of observations and their summarized temporal characteristics will be used to determine whether different types of trajectories emerge. Hierarchical cluster analysis will label patients for each of the cluster solutions and the usefulness of patient labelling will be evaluated by their predicted gait performance. The extracted patient type will be included in random forests or boosting to evaluate its importance. The extracted patient type could also be used jointly with other predictors suggested as important in either a linear/logistic (mixed) model or an extended cox proportional hazard model, which are more traditional statistical approaches. While predictive performance remains the key goal, such models would be more interpretable on the potential underlying mechanism, with parameter estimates and confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Hospitalized at the Neurology ward of UZ Brussel
* Diagnosed with first-ever stroke (as defined by the World Health Organisation)
* Able to provide written or verbal informed consent

Exclusion Criteria:

* Other neurological or orthopaedic problems leading to impaired gait
* Severe deficits of communication, memory or understanding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute stroke survivors
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulation Categories | Change over time between baseline (≤ 3 days post-stroke), discharge (anticipated average of 10 days post-stroke) and 3 months follow-up
  The Functional Ambulation Categories (FAC) will be used to measure walking ability in patients assigned to cohort 1. The score ranges from 0-5, with a higher score reflecting towards a more independent walking ability.
6-minutes walking test | Change over time between baseline (≤ 3 days post-stroke), discharge (anticipated average of 10 days post-stroke) and 3 months follow-up
  The 6-minutes walking test (6MWT) will evaluate the walking endurance of the subjects in cohort 2. During this test we will measure the distance walked over a span of 6 minutes.

SECONDARY OUTCOMES:
Rivermead Mobility Index | Baseline (≤ 3 days post-stroke), discharge (anticipated average 10 days post-stroke), 3 months
  The Rivermead Mobility Index (RMI) will assess functional mobility in gait, balance and transfers in subjects of cohort 1. The RMI consists of 14 self-reported items and 1 direct observation with an overall maximum score of 15 points. A higher score represents a better outcome.
Gait speed | Baseline (≤ 3 days post-stroke), discharge (anticipated average 10 days post-stroke), 3 months
  Gait speed (m/s) will be evaluated by using wearable motion sensors (Gait Up) during the 6MWT in patients assigned to cohort 2.
Oxygen cost | Baseline (≤ 3 days post-stroke), discharge (anticipated average 10 days post-stroke), 3 months
  Oxygen cost (ml/kg/m) will be observed by respiratory gas analysis with the MetaMax 3B. All subjects from cohort 2 will wear this system during their 6MWT.
Muscle strength | Baseline (≤ 3 days post-stroke), 3 days after baseline assessment, discharge (anticipated average 10 days post-stroke), 3 months
  Muscle strength of the lower extremities will be assessed on one hand with the Motricity Index, a clinical tool which measures strength in the ankle dorsiflexors, knee extensors and hip flexors. On the other hand, we will use a hand-held dynamometer (MicroFET2) to assess the maximal isometric muscle strength of the knee extensors and ankle dorsiflexors (Newton) on the paretic and non-paretic side.
Grip strength | Baseline (≤ 3 days post-stroke), 3 days after baseline assessment, discharge (anticipated average 10 days post-stroke), 3 months
  Maximal hand grip strength will be assessed with the Martin Vigorimeter (KPa) on both sides.
Muscle Fatigue | Baseline (≤ 3 days post-stroke), 3 days after baseline assessment, discharge (anticipated average 10 days post-stroke), 3 months
  To observe muscle fatigue, we will use the Martin Vigorimeter. Muscle fatigue is defined as the time during which handgrip strength drops to 50% of its maximal value during sustained maximal contraction.
Muscle Mass | Baseline (≤ 3 days post-stroke), 3 days after baseline assessment, discharge (anticipated average 10 days post-stroke), 3 months
  A bioelectrical impedance analysis (BIA) system will be used to assess the muscle mass of the subjects.
Muscle architecture | Baseline (≤ 3 days post-stroke), 3 days after baseline assessment, discharge (anticipated average 10 days post-stroke), 3 months
  We will use ultrasound technique to evaluate the muscle architecture of the m. tibialis anterior and the m. gastrocnemius medialis. The architectural qualities of the muscles involve: muscle thickness, pennation angle, fascicle length and cross-sectional area.
Muscle Tone | Baseline (≤ 3 days post-stroke), 3 days after baseline assessment, discharge (anticipated average 10 days post-stroke), 3 months
  The Modified Ashworth Scale (MAS) will evaluate the amount of spasticity on both sides in the m. quadriceps, m. gastrocnemius and m. soleus based on a 6-point ordinal scale, with a higher score reflecting towards more spasticity in the muscle.
Circulating biomarkers | Baseline (≤ 3 days post-stroke), 3 days after baseline assessment, discharge (anticipated average 10 days post-stroke), 3 months
  Through blood sampling we investigate following circulating biomarkers: Brain-derived neurotrophic Factor (BDNF), inflammation related biomarkers (CRP, IL1β, TNFα, IL1ra, IL6, IL-8, IL-10, IL-15), heat shock proteins (hsp) (hsp27 and hsp 70) and Irisin.
Short Physical Performance Battery | Baseline (≤ 3 days post-stroke), 3 days after baseline assessment, discharge (anticipated average 10 days post-stroke), 3 months
  The Short Physical Performance Battery (SPPB) will be used to evaluate balance and mobility of the subjects. It is a test which combines the results of a gait speed test, a balance test and a chair stand test.
Fatigue Assessment Scale | Baseline (≤ 3 days post-stroke), 3 days after baseline assessment, discharge (anticipated average 10 days post-stroke), 3 months
  The Fatigue Assessment Scale (FAS) will be used to assess physical and mental fatigue. The questionnaire consists of 10 statements which have to be answered with one out of five categories varying from never to always.

CONTACTS AND LOCATIONS:
Overall Officials: David Beckwée, Prof. Ph.D, Study Chair — Vrije Universiteit Brussel; Eva Swinnen, Prof. Ph.D, Study Chair — Vrije Universiteit Brussel; Lotte Cuypers, Dra., Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium